CLINICAL TRIAL: NCT05946681
Title: Sildenafil Citrate to Improve Maternal and Neonatal Outcomes in Low-resource Settings
Acronym: PRISM
Status: Completed | Type: Observational
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Global Network for Women's and Children's Health Research (Other); University of Alabama at Birmingham (Other); University Teaching Hospital, Lusaka, Zambia (Other); RTI International (Other)
Responsible Party: Sponsor
Other Study IDs: GN03 PRISM Sildenafil Pilot
Record Dates: First submitted 2023-06-14; First posted 2023-07-14 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2023-11

CONDITIONS: Fetal Distress; Perinatal Asphyxia; Birth Asphyxia; Stillbirth
Keywords: Fetal Distress; Perinatal Asphyxia; Sildenafil Citrate; Fetal Heart Rate Monitoring; Zambia
MeSH Terms: conditions — Fetal Distress; Asphyxia Neonatorum; Stillbirth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PRISM pilot feasibility study consists of two phases to determine: 1) to delivery practices, rates of primary and secondary outcomes, and feasibility of enrollment rates, and 2) to assess the feasibility and acceptability of the intervention and expected enrollment rates, and estimate the effect size of sildenafil citrate on maternal and neonatal outcomes in a low resource settings in preparation for the main RCT.

DETAILED DESCRIPTION:
The primary objectives of the PRISM pilot study relate to feasibility of a large randomized controlled trial of intrapartum sildenafil citrate and will aid in design of a definitive trial among pregnant women to day 42 postpartum (pp) and their newborns to day 28 pp. The pilot will help prepare for the main trial by allowing the investigators to:

* Determine the rate and indication for fetal heart rate monitoring practices;
* Determine the rate and indications for operative delivery;
* Inform the rates of relevant primary and secondary outcomes to possibly target in a large randomized controlled trial of intrapartum sildenafil citrate;
* Assess the feasibility and acceptability of the intervention and expected enrollment rates;
* Estimate the effect size of sildenafil citrate on maternal and neonatal outcomes in a low resource setting.

ELIGIBILITY:
Inclusion Criteria:

* Admission to facility with plan for spontaneous or induced vaginal delivery
* Early stage of labor (≤ 6 cm cervical dilation per local standard) at ≥ 37 weeks gestation
* Age ≥ 18 years of age
* Presence of single live fetus confirmed via a fetal heart rate by Doptone in cephalic position
* Provision of written informed consent [Note: if written consent is obtained at an early time, verbal re-confirmation is required at time of enrollment]

Exclusion Criteria:

* Non-emancipated minors (as per local regulations)
* Plan for Cesarean delivery or history of cesarean section prior to enrollment*
* Unknown gestational age
* Advanced stage of labor (>6 cm or 10 cm cervical dilation per local standards) and pushing or too distressed to understand, confirm, or give informed consent regardless of cervical dilation
* Not capable of giving consent due to other health problems such as obstetric emergencies (for example, antepartum hemorrhage) or mental disorder;
* Any medical condition considered a contraindication, including contraindication to sildenafil therapy, per the judgement of site investigators
* Any maternal medical condition or status that precludes informed consent
* Recognized fetal anomaly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women who are delivering in a participating health facility will be screened for eligibility
Study Population: The pilot observational study will be undertaken in two sites in Zambia; one in a Level 3 delivery facility and a Level 2 delivery facility in Lusaka. A maximum of 1000 women per site will be enrolled in the pilot study. Each site will prospectively collect up to six months of data, three months of piloting forms and non-drug interventions. A subsequent small RCT with study medication will enroll 500 participants over a period of up to three months per site. Enrollment will take place in pre-identified health facilities where women present for labor and delivery.
Sampling Method: Non-Probability Sample
Enrollment: 1017 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Effect size estimate of the intervention on the incidence of the composite neonatal outcome. | From delivery to 7 days post delivery
  The outcome will be measured by overall number of eligible consented participants and incidence of the composite neonatal outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Elwyn Chomba, MD, Principal Investigator — Levy Mwanawasa Medical University
Locations (1):
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes